CLINICAL TRIAL: NCT00824967
Title: Not Pharmacologic Treatment Has Illness of Alzheimer and Pathologies Related. Application in Disturbances of Behaviour in EHPAD
Brief Title: Non Pharmacological Management of Behavioural Symptoms in Nursing Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 07-PP-03
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2009-01

CONDITIONS: ALZHEIMER Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- The reference group (No Intervention): one will take care of the patient in a habitual way: no consultation additional, step of exam on top of that...
- 2- The intervention group (Other): Training and valuation of the treating personnel
  Interventions: Other: Training and valuation of the treating personnel

INTERVENTIONS:
Other: Training and valuation of the treating personnel — Training and valuation of the treating personnel
  Arms: 2- The intervention group

SUMMARY:
Background: Behavioural and psychological symptoms of dementia (BPSD) are often reported in institutions for the elderly.

Objective: To evaluate the effectiveness of a staff education intervention to manage BPSD in older people with a diagnosis of dementia.

DETAILED DESCRIPTION:
Background: Behavioural and psychological symptoms of dementia (BPSD) are often reported in institutions for the elderly.

Objective: To evaluate the effectiveness of a staff education intervention to manage BPSD in older people with a diagnosis of dementia.

Methods: The trial was conducted in 16 nursing homes; 306 patients with a diagnosis of dementia and presenting BPSD were selected. Nursing homes were randomly allocated to an intervention group or a control group. An eight-week staff education and training programme was conducted in the nursing homes in the intervention group. The main outcome measures were the Cohen-Mansfield Agitation Inventory (CMAI) and an observation scale score. Assessments were done at baseline (W0), at the end of the 'intervention' period (W8) and 12 weeks after (W20).

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer disease

Exclusion Criteria:

* Not alzheimer disease

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Changes at the behavioural assessment (CMAI, OS, NPI) after 8 weeks of intervention | 8 weeks after intervention

SECONDARY OUTCOMES:
Changes at the behavioural assessment (CMAI, OS, NPI) 16 weeks after the end of the intervention | 16 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PhD, Principal Investigator — CHU de Nice - CM2R - Hôpital de Cimiez - 4 avenue reine victoria - 06 003 Nice cedex 1
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria, Nice, Alpes-Maritimes, France